CLINICAL TRIAL: NCT01666743
Title: A Multicenter Study to Describe the Safety and Efficacy of Ceftaroline Fosamil in Elderly Subjects With Community-Acquired Bacterial Pneumonia
Brief Title: Safety and Efficacy Study of Ceftaroline in Elderly Subjects With Community-Acquired Bacterial Pneumonia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in strategy.
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPT-MD-34
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Community-Acquired Bacterial Pneumonia (CABP)
Keywords: Community-Acquired Pneumonia; Lung; Adult; Infections
MeSH Terms: conditions — Community-Acquired Pneumonia; Infections | interventions — Ceftaroline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ceftaroline fosamil (Experimental): IV ceftaroline fosamil 600 mg infused over 60 (± 10) minutes every 12 hours (dosing may be adjusted for renal impairment)
  Interventions: Drug: Ceftaroline fosamil

INTERVENTIONS:
Drug: Ceftaroline fosamil — IV ceftaroline fosamil 600 mg infused over 60 (± 10) minutes every 12 hours (dosing may be adjusted for renal impairment)
  Other Names: Teflaro®; PPI-0903; TAK-599; TAK599; PPI0903

SUMMARY:
The purpose of this study is to determine the safety and efficacy of ceftaroline fosamil in elderly subjects with community-acquired bacterial pneumonia (CABP) receiving antibiotic therapy in the hospital.

DETAILED DESCRIPTION:
This is a multicenter study of ceftaroline fosamil in elderly subjects (≥ 65 years of age) with CABP. Adjunctive macrolide therapy is to be used at the Investigator's discretion. A switch to oral treatment may be allowed at the discretion of the Investigator. The total duration of therapy is 5 to 7 days; a minimum of 48 hours of study drug is required.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 65 years of age.
2. Presence of CABP warranting hospitalization.
3. Acute illness with ≥ 2 clinical signs or symptoms of lower respiratory tract infection.
4. Radiographically confirmed pneumonia.

Exclusion Criteria:

1. History of any hypersensitivity or allergic reaction to any β-lactam or macrolide antibacterial agent.
2. Confirmed or suspected respiratory tract infection due solely to an atypical bacterial, mycobacterial, viral, or fungal pathogen.
3. More than 24 hours of potentially effective antibacterial therapy within 96 hours prior to enrollment.
4. Life expectancy of < 30 days or presence of an order of Do Not Resuscitate (DNR).
5. Evidence of significant hematologic, hepatic, or immunologic impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of ceftaroline fosamil in elderly subjects (≥ 65 years) with community-acquired bacterial pneumonia (CABP) | Between 3 and 33-37 days
  Safety evaluations will be conducted and assessments will include:
  * Adverse events including deaths will be evaluated.
  * Laboratory: complete blood count with differential, and chemistry panel.

SECONDARY OUTCOMES:
Evaluate the efficacy of ceftaroline fosamil in elderly subjects (≥ 65 years) with community-acquired bacterial pneumonia (CABP) | 30 days following discharge from the hospital, anticipated between 33 to 37 days.
  Efficacy outcome measures:
  * Time to clinical stability
  * Length of stay
  * Clinical outcome at End-of-Intravenous Study Drug, End-of-Therapy, and Test-of-Cure
  * Mortality
  * 30-day readmission

REFERENCES:
- See also: Sponsor Website — http://www.cerexa.com